CLINICAL TRIAL: NCT00556634
Title: Randomized, Double-Blinded Clinical Trial to Evaluate the Incidence and Severity of Neuropsychiatric Side Effects and Antiviral Efficacy of Efavirenz Given as a Stepped Dosage Over 2 Weeks Versus the Usual Dosage in HIV-Infected Patients.
Brief Title: Incidence and Severity of Neuropsychiatric Adverse Events of Efavirenz Given as a Stepped Dosage vs. the Usual Dosage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Luis Fernando Lopez-Cortes, Servicio Andaluz de Salud. Hospitales Uiversitarios Virgen del Rocíoi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAEI_EFV
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: HIV-1 Infection; HIV Infection
Keywords: HIV; efavirenz; central nervous system; adverse effects
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator)
  Interventions: Drug: Efavirenz
- A (Experimental)
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — Efavirenz given in a stepped dosage over 2 weeks (200 mg qd for 6 days plus placebo, 400 mg qd for 7 days plus placebo and 600 mg qd from day 14 forward)
  OR
  Efavirenz usual dosage (600 mg/day from the first day)

SUMMARY:
Background: Neuropsychiatric side effects (NPSEs) occur in a significant proportion of subjects after initiation of efavirenz (EFV) and may limit its use in certain patients.

Objectives: To evaluate the incidence and severity of NPSEs and antiviral efficacy of EFV given as a stepped dosage over 2 weeks versus the usual dosage.

Methods: Randomized, double blind, multicentric clinical trial in which a progressive dosage (arm A: 200 mg qd for 6 days, 400 mg qd for 7 days and 600 mg qd from day 14 forward) was compared with conventional administration (arm B: 600 mg qd from the first day). All patients received additional treatment with 2 NRTIs.

The incidence and intensity of NPSEs and sleep disorders were assessed using a Likert-type scale specifically designed. Efficacy was assessed by percent of virological failures.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* HIV-1 infection
* Women of child-bearing age: negative pregnancy test
* Ability to understand and sign a written consent form

Exclusion Criteria:

* Pregnancy..
* Illegal drug or methadone use.
* Major psychiatric disease antecedents or starting new psychotropic agents in the last 4 weeks
* Concomitant treatment with rifamycins, protease inhibitors or drugs which interfere the pharmacokinetic of efavirenz.
* Hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
incidence and severity of neuropsychiatric side effects | 4 weeks

SECONDARY OUTCOMES:
Virological efficacy | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD, Study Director — Hospitales Universitarios Virgen del Rocio. Seville. Spain
Locations (10):
- Spain (10):
  - Hospital Torrecardenas, Almería, Almeria
  - Hospital Universitario Puerta del Mar, Cadiz, Cadiz
  - Hospital de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba, Cordoba
  - Hospital Juan Ramon Jimenez, Huelva, Huelva
  - Hospital Universitario Carlos Haya, Málaga, Malaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospitales Universitarios Virgen del Rocio, Seville, Seville
  - Hospital Universitario de Valme, Seville, Seville
  - Hospital Universitario Virgen Macarena, Seville, Seville

REFERENCES:
- [Derived] Gutierrez-Valencia A, Viciana P, Palacios R, Ruiz-Valderas R, Lozano F, Terron A, Rivero A, Lopez-Cortes LF; Sociedad Andaluza de Enfermedades Infecciosas. Stepped-dose versus full-dose efavirenz for HIV infection and neuropsychiatric adverse events: a randomized trial. Ann Intern Med. 2009 Aug 4;151(3):149-56. doi: 10.7326/0003-4819-151-3-200908040-00127. Epub 2009 Jul 6. PMID 19581631